CLINICAL TRIAL: NCT02583932
Title: Randomized Controlled Trial of the Meaning-Making Intervention (MMi) In People Newly Diagnosed With Advanced Cancer: Full Trial
Brief Title: Randomized Controlled Trial of the Meaning-Making Intervention (MMi) In Newly Diagnosed Advanced Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jewish General Hospital (Other)
Collaborators: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Melissa Henry, Clinician-Scientist, Jewish General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: MM-JGH-15-100
Record Dates: First submitted 2015-10-16; First posted 2015-10-22 (Estimated); Last update posted 2021-01-08 (Actual); Status verified 2021-01

CONDITIONS: Advanced Cancer
Keywords: Randomized controlled trial; Psychological; Meaning; Existential; Quality of life; Intervention; Cancer; Advanced disease; New diagnosis
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Masking Description: Investigators and care providers are masked as to group assignment
Oversight: Data Monitoring Committee: No

ARMS (3):
- Meaning-Making intervention (MMi) (Experimental): The MMi is a brief, individualized and manualized therapeutic approach based on post-trauma literature and designed to facilitate a search for meaning following a cancer diagnosis. The MMi consists of 3-4 weekly sessions of 30-90 min each with an intervener (psychologist, social worker, or nurse) who provides the necessary ingredients to foster a good therapeutic alliance (i.e., trust, warmth, empathy, neutrality, and authenticity), encourages self-exploration and systematically addresses different levels of meaning (i.e., situational, global, existential, historical).
  Interventions: Drug: Meaning-Making intervention (MMi)
- Empathic Visitor (EV) (Placebo Comparator): Empathic visitors will meet with patients over 3-4 weekly sessions of 30-90 minutes as in the experimental group. They will provide the basic ingredients for fostering a good therapeutic relationship (i.e., trust, warmth, empathy, neutrality and authenticity) without further intervention or probing. The empathic listener will be specifically instructed to avoid initiating discussions about meaning (e.g., perspective-taking, how the patient interprets his/her feelings and thoughts, understands his/her illness and meaning in life), and focus discussions on what is currently happening (rather than on the interface between past and present). If the patient initiates discussions about these topics, the visitor will simply listen without further intervening.
  Interventions: Behavioral: Empathic Visitor
- Usual Care Control Group (No Intervention): Treatment as usual in tertiary care hospital, typically medically-focused. All participants will be free to use hospital- or community-based supports, which will be tracked in all groups throughout the study by questionnaire and through a chart review. Both recruiting centres include well established psychosocial oncology services including psychiatrists, psychologists and social workers.

INTERVENTIONS:
Drug: Meaning-Making intervention (MMi) — The MMi is a brief, individualized and manualized therapeutic approach based on post-trauma literature and designed to facilitate a search for meaning following a cancer diagnosis.
  Other Names: MMi
  Arms: Meaning-Making intervention (MMi)
Behavioral: Empathic Visitor — They will provide the basic ingredients for fostering a good therapeutic relationship (i.e., trust, warmth, empathy, neutrality and authenticity) without further intervention or probing.
  Other Names: Attention-Control
  Arms: Empathic Visitor (EV)

SUMMARY:
To test whether the Meaning-Making intervention (MMi)(Lee, 2004) plus usual care increases the sense of meaning in life in people newly diagnosed with any type of advanced cancer, compared to similar people who receive 1) usual care alone or 2) usual care plus visits from an empathic visitor, at 2 months after randomization to one of these treatments. The investigators will also evaluate whether any effect is present at 4 and 6 months post-randomization, and the MMi's impact on anxiety/depression, quality of life, existential wellbeing, and posttraumatic growth. To answer our research questions 471 newly diagnosed (<6 months) advanced cancer patients (stages III or IV) will be studied.

DETAILED DESCRIPTION:
Background: Psychosocial interventions are effective for all types of cancer in preventing and addressing distress and enhancing quality of life. However, most neglect existential issues. Issues of meaning and meaninglessness are especially important existential concerns for advanced cancer patients and crucial in determining their quality of life. Adaptation can be promoted and current and/or future existential crises curtailed by an early, psychologically growth-promoting intervention such as the Meaning-Making intervention (MMi)(Lee, 2006), helping patients adapt more quickly or fully, and preparing them for stormy periods ahead such as the end of life. However, it is not known whether: 1) the MMi can help patients newly diagnosed with advanced cancer; 2) it increases a sense of meaning in life; 3) its impact lasts beyond the end of the intervention; and 4) the effect shown is due to the MMi or a similar effect could be obtained by having someone listen empathically for the same amount of time as it takes to administer the MMi.

The investigators now want to test its efficacy in a full 3-arm randomized controlled trial for newly diagnosed advanced cancer patients. They will roll in the feasibility pilot study data (n=60) since it demonstrated that the initial protocol was feasible and the investigators therefore did not view or analyze the outcome data (it was viewed only by the research coordinator) and the design stayed the same (ClinicalTrials.gov Identifier: NCT01693991). .

Primary Hypothesis: Adding the MMi to usual care (experimental group) enhances meaning in life on the FACIT-Sp-12 meaning subscale among newly diagnosed advanced cancer patients, compared with those receiving usual care plus meetings with an empathic non-professional visitor (i.e., attention-control group) or usual care alone, at 2 months post-randomization. "Meaning in life" (primary outcome) is defined as the belief that one's life has significance and purpose (i.e., global meaning) and "newly diagnosed advanced cancer patient" is defined as the 6 months after first occurrence of, progression to, or recurrence of stage III or IV cancer.

Secondary hypotheses: The Experimental Group will have decreased anxiety and depression (Hospital Anxiety and Depression Scale), increased overall quality of life (McGill Quality of Life Questionnaire (MQOL) Total), existential wellbeing (MQOL Existential Wellbeing), and posttraumatic growth (Post-Traumatic Growth Inventory), compared to the Attention-Control and Usual Care groups at 2 months post-randomization. Furthermore, the MMi effects are present at 4 and 6 months post-randomization. Additional analyses: The investigators plan subgroup analyses of effect modifiers such as gender, degree of baseline perceived life-threat, initial level of psychological distress, initial level of meaning in life, and degree of experienced physical wellbeing.

Design and method: RCT with 471 newly diagnosed advanced cancer patients assigned randomly to the Experimental Group, Attention-Control, or Usual Care. Patients will complete self-report questionnaires measuring outcomes at baseline, 2, 4 and 6 months post-randomization.

Significance of the research: Advanced cancer patients are confronted with the possibility of imminent death and consequently struggle to search for meaning in their plight. An early, psychologically growth-promoting intervention is especially important for these patients to prevent further distress within a lifespan that is likely to be limited. Interventions designed to promote psychological wellbeing and enhance quality of life usually fail to address this important existential dimension and pathway to improved wellbeing. The MMi offers a promising avenue to help advanced cancer patients adjust to their diagnosis and improve their quality of life, helping them to adapt more quickly or fully. If the results of this RCT are positive, focus groups and interviews with key stakeholders indicate that it will be integrated into routine cancer care, with outreach activities designed to equip the oncology healthcare community to address meaning and existential issues in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with advanced cancer (stage III or IV --TNM classification system); first occurrence, progression or recurrence of any type of solid tumour <4 months at referral and <4 months at randomization, as well as Hodgkin's and non-Hodgkin's lymphoma
2. Physically able (referring clinician- and self-perceived) and willing to participate in weekly MMi or attention control sessions.
3. >18 years old.
4. Alert and capable of giving free and informed consent according to the referring clinician.
5. Able to speak and read English or French.

Exclusion Criteria:

1. Karnofsky Performance Status (KPS) score <60 (rated by referring oncologists/nurses or Research Coordinator) or expected survival <6 months according to clinical judgment of physicians and/or nurses.
2. Currently experiencing severe radiotherapy side-effects. These patients will only be included in the study when they will have recovered from these severe side-effects and when they feel they can participate in the study. Severe radiotherapy side-effects are defined as a score of 3 or 4 on any of the site-specific toxicity markers of the Eastern Cooperative Oncology Group (ECOG) Common Toxicity Criteria or with > 3 markers with a score of 2, as evaluated by the treating physician (in consultation with the radiotherapist).
3. Currently suicidal (present a score ≥2 on the Beck Depression Inventory suicide item, or self-reported chronic suicidal ideations in the pre-cancer diagnosis period, assessed by the Research Coordinator or Research Assistant (RA) during the consent meeting.
4. Known diagnosis of schizophrenia or schizoaffective disorder.
5. Planning a trip within 2 months that would interrupt intervention delivery.
6. Current or former therapy with Dr. Henry (the PI who already does meaning-based interventions at the Jewish General Hospital).
7. Attending or planning to attend either of the MUHC CanSupport workshops entitled " You are stronger than you think" or "Vous êtes plus fort que vous ne le pensez: Donnez un sens au cancer".
8. Previously receiving any version of the "Reflections Workbook : A self care guide to understanding the experience of cancer".

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 179 (Actual)
Dates: Start 2015-10; Primary Completion 2020-08 (Actual); Study Completion 2020-08 (Actual)

PRIMARY OUTCOMES:
Meaning in life measured by Facit-Sp-12 meaning subscale | 2 months post-randomization
  Facit-Sp-12 meaning subscale

SECONDARY OUTCOMES:
Existential Wellbeing measured by McGill Quality of Life (MQOL) Existential Wellbeing subscale | 2 months post-randomization
  McGill Quality of Life (MQOL) Existential Wellbeing subscale
Anxiety and depression measured by Hospital Anxiety and Depression Scale (HADS) Total score | 2 months post-randomization
  Hospital Anxiety and Depression Scale (HADS) Total score
Quality of life measured by McGill Quality of Life (MQOL) Total score | 2 months post-randomization
Post-traumatic growth measured by Post-Traumatic Growth Inventory (PTGI) Total score | 2 months post-randomization
  Post-Traumatic Growth Inventory (PTGI) Total score

OTHER OUTCOMES:
All of the abovementioned outcomes | 4 and 6 months post-randomization
  Exploratory analyses

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Henry, Ph.D., Principal Investigator — Jewish General Hospital; Robin Cohen, Ph.D., Principal Investigator — Jewish General Hospital
Locations (2):
- Canada (2):
  - Jewish General Hospital, Montreal, Quebec
  - McGill University Health Centre (MUHC), Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No